CLINICAL TRIAL: NCT02478164
Title: Phase II Trial of Ponatinib in Patients With Bevacizumab-Refractory Glioblastoma
Brief Title: Trial of Ponatinib in Patients With Bevacizumab-Refractory Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Eudocia Quant Lee, MD, Eudocia Lee, MD, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-163
Record Dates: First submitted 2015-06-12; First posted 2015-06-23 (Estimated); Results first posted 2018-04-02 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-06

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — ponatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ponatinib (Experimental): Drug will be administered once daily per cycle through oral ingestion.
  Interventions: Drug: Ponatinib

INTERVENTIONS:
Drug: Ponatinib
  Other Names: ponatinib hydrochloride; Iclusig

SUMMARY:
This research study is studying a chemotherapy as a possible treatment for recurrent glioblastoma that has not responded to bevacizumab. The name of the study drug involved in this study is Ponatinib.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved Ponatinib for your specific disease but it has been approved for other uses.

Ponatinib is a drug that may stop cancer cells from growing by affecting different kinds of proteins in cancer cells. Glioblastoma cells can be driven by mutated forms of a protein called c-kit (KIT) which are present in glioblastoma cells. Laboratory studies suggest that ponatinib has activity against mutated forms of (KIT) which is important in glioblastoma and therefore suggests that ponatinib may help to control the growth of glioblastoma. In this research study the study team is looking to see if ponatinib is safe and is able to control the growth of glioblastoma in people who have not responded to treatment with bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Karnofsky performance status ≥ 60
* Participants must have histologically confirmed glioblastoma or variants. Subjects with initial diagnosis of a lower grade glioma are eligible if a subsequent biopsy is determined to be glioblastoma or variants.
* Patients must have an unequivocal progression by magnetic resonance imaging (MRI) or computed tomography (CT) scan. A scan must be performed within 14 days prior to registration and on a steroid dose that has been stable or decreasing for at least 5 days. If the steroid dose is increased between the date of imaging and initiation of study treatment, a new baseline MRI/CT is required.
* Participants must have bi-dimensionally measurable disease with a minimum measurement of 1 cm per dimension on MRI performed within 14 days prior to first treatment. If receiving corticosteroids, participants must be on a stable or decreasing dose of corticosteroids for at least 5 days prior to baseline MRI.
* There is no limit on the number of prior relapses but the most recent relapse must be the first relapse on a bevacizumab-containing regimen.
* Participants must have normal organ and marrow function as defined below:

  * Leukocytes ≥3,000/mcL (≥ 3,000/mm3)
  * Absolute neutrophil count ≥ 1,500/mcL (> 1,500/mm3)
  * Platelets ≥ 100,000/mcL (≥ 100,000/ mm3)
  * Total bilirubin ≤ 1.5 X institutional upper limit of normal, unless due to Gilbert's syndrome.
  * AST (SGOT)/ALT (SGPT) ≤ 2.5 X institutional upper limit of normal
  * Serum Creatinine ≤ 1.5 X institutional upper limit of normal or or creatinine clearance > 60 mL/min/1.73 m2 (per 24 hour urine collection or calculated according to the Cockcroft-Gault formula) for subjects with creatinine levels above the institutional normal
  * Serum lipase and amylase ≤ 1.5 X institutional upper limit of normal.
* Participants must have fully recovered (grade ≤ 1 or baseline or deemed irreversible) from any clinically significant acute toxicity related to prior therapy (with the exception of lymphopenia, which is common after therapy with temozolomide). Patients who discontinued bevacizumab previously due to a bevacizumab-related toxicity will not be allowed to participate.
* The following time periods must have elapsed prior to the planned start date of study treatment:

  * ≥2 weeks or 6 half lives from any approved TKIs or investigational agent, whichever is longer
  * ≥4 weeks from prior cytotoxic therapy, except ≥ 3 weeks from last dose of temozolomide and ≥6 weeks from nitrosoureas or mitomycin C
  * ≥2 weeks from non-cytotoxic agents
  * ≥ 3 weeks from bevacizumab
* Participants must have developed progressive disease after receiving prior radiation therapy and must have an interval of at least 12 weeks from the completion of any radiation therapy to study entry (unless progressive tumor growth is outside the radiation field or there is histopathological confirmation of recurrent tumor).
* Participants may not have received prior therapy with any other Src, PDGFR, or FGFR inhibitor. Prior treatment with an anti-VEGFR or anti-VEGF agent is also allowed but only one relapse following a bevacizumab-containing regimen is allowed.
* For females of childbearing potential, a negative serum pregnancy test must be documented prior to registration.

  --- NOTE: In addition to screening, serum pregnancy test must be performed on females of childbearing potential within 72 hours before the start of investigational product. When possible, these tests can be one-in-the-same (if screening pregnancy test was performed within 72 hours of first ponatinib dose, no need to repeat).
* The effects of ponatinib on the developing human fetus are unknown. For this reason and because ponatinib is known to be teratogenic in animal models, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and through 4 months after the end of treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

NOTE: Consent documents can be signed up to 30 days prior to registration. If >30 days has elapsed since patient signed the consent document, s/he must re-consent (new signature) before proceeding to register onto study.

* Participants must have sufficient tissue from prior surgery for confirmation of diagnosis and correlative studies. The following amount of tissue is required:

  * 15 (5 μm thick) unstained formalin fixed paraffin embedded (FFPE) sections
  * 1-2 H&E stained slides, or additional unstained 5 μm slide(s) for staining
* Protocol treatment plan must include beginning therapy within 5 consecutive days after registration.

Exclusion Criteria:

* Participants may not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ponatinib.
* Participants who have received prior treatment with interstitial brachytherapy, stereotactic radiosurgery, or implanted chemotherapy sources, such as wafers of polifeprosan 20 with carmustine
* Participants with poorly controlled diabetes defined as a HgbA1c ≥ 7.0%
* Participants with grade ≥ 3 peripheral motor or sensory neuropathy.
* Participants receiving any medications or substances that are moderate and strong inhibitors or inducers of CYP3A4, including enzyme-inducing anti-epileptic drugs (EIAEDs) within 14 days before the first dose of ponatinib will be excluded. This category includes phenobarbital, phenytoin, fosphenytoin, primidone, carbamazepine, and oxcarbazepine. Lists including medications and substances known or with the potential to interact with CYP3A4 isoenzymes are provided in Appendix B.

  --- NOTE: Participants must avoid consumption of Seville orange (and juice), grapefruit or grapefruit juice, grapefruit hybrids, pummelos and exotic citrus fruits from 7 days prior to the first dose of study drug and during the entire study treatment period due to potential CYP3A4 interaction.
* Participants taking medications that are known to be associated with Torsades de Pointes or QT prolongation. Refer to Tables C-1 and C-2 of Appendix C for a list of prohibited drugs.
* Participants cannot take any herbal preparations/medications on study or within 7 days prior to first dose of study drug, including but not limited to: St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, ginseng.
* Participants who underwent major surgery (including craniotomy) or significant traumatic injury within 28 days prior to initiating therapy. Baseline MRIs for participants who underwent salvage surgery must be obtained at least 4 weeks after procedure and there must be measurable disease.
* Participants who underwent minor surgical procedure within 7 days prior to initiating therapy.
* History of a bleeding disorder.
* Patients with gastrointestinal bleeding or any other hemorrhage/bleeding event CTCAE Grade >/= 3 within 30 days prior to study entry.
* Patients whose MRI scan demonstrates intratumoral hemorrhage or peritumoral hemorrhage are not eligible for treatment if deemed significant by the treating physician. If there are questions, the treating physician should contact the study's Overall PI, Dr. Lee
* History of acute pancreatitis within 1 year of study treatment or a history of chronic pancreatitis.
* History of alcohol abuse.
* Uncontrolled hypertriglyceridemia (triglycerides >450 mg/dL)
* Clinically significant, uncontrolled, or active cardiovascular disease, specifically including, but not restricted to:

  * Any history of myocardial infarction
  * Any history of clinically significant (as determined by the treating physician) atrial arrhythmia
  * Any history of ventricular arrhythmia
  * Any history of Cerebrovascular accident or transient ischemic attack (TIA)
  * Any history of peripheral arterial occlusive disease requiring rvascularization
  * Unstable angina within 6 months prior to enrollment
  * Congestive heart failure within 6 months prior to enrollment
  * Venous thromboembolism including deep venous thrombosis or pulmonary embolism within 6 months prior to enrollment
  * Unacceptable Screening Baseline Cardiovascular Assessment:

    * Baseline MUGA or Echocardiogram demonstrating LVEF < 50 %
    * QTc > 480 msec on screening ECG (using the QTcF formula)
* Uncontrolled hypertension (diastolic blood pressure >90 mm Hg; systolic >140 mm Hg). Patients with hypertension should be under treatment on study entry to effect blood pressure control.
* Ongoing or active infection. The requirement for intravenous (IV) antibiotics is considered active infection.
* Known history of human immunodeficiency virus (HIV). Testing is not required in the absence of prior documentation or known history.
* Pregnant or breastfeeding.

  -- Pregnant women are excluded from this study because ponatinib has potential for teratogenic or abortifacient effects in animal models. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with ponatinib, breastfeeding should be discontinued if the mother is treated with ponatinib. These potential risks may also apply to other agents used in this study.
* Malabsorption syndrome or other gastrointestinal illness that could affect oral absorption of study drugs.
* Individuals with a history of a different malignancy, other than cervical cancer in situ, basal cell or squamous cell carcinoma of the skin, are ineligible, except if they have been disease-free for at least 5 years, and are deemed by the investigator to be at low risk for recurrence of that malignancy OR if the other primary malignancy is neither currently clinically significant nor requiring active intervention.
* Any condition or illness that, in the opinion of the Investigator, would compromise patient safety or interfere with the evaluation of the drug.
* HIV-positive individuals on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with ponatinib. In addition, these individuals are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-07-13 (Actual); Primary Completion 2017-07-08 (Actual); Study Completion 2018-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eudocia Lee, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study began enrolling on 7/13/2015 and enrolled the last participant on 6/13/2017. Enrollment was stopped during a planned interim analysis due to futility. 17 participants were enrolled, but only 15 went on to receive ponatinib study treatment, as 2 participants withdrew after enrolling and before beginning ponatinib.
Period: Overall Study
Arm/Group | Ponatinib
Started | 15 (17 participants enrolled. 15 of 17 received ponatinib as 2 participants withdrew prior to ponatinib.)
Completed | 0
Not Completed | 15
Not completed — Lack of Efficacy | 13
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ponatinib
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 62 [28 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 1
  Unknown or Not Reported | 0
Initial Glioma Diagnosis [Count of Participants; unit: Participants]
  Anaplastic Oligodendroglioma | 1
  Astrocytoma | 1
  Oligodendroglioma | 1
  Glioblastoma Multiforme | 12
Current Tumor Diagnosis [Count of Participants; unit: Participants] | 15
Number of Prior Relapses [Count of Participants; unit: Participants]
  Second relapse | 10
  Third relapse | 4
  Fourth relapse | 1
  First relapse | 0
Baseline Karnofsky performance status (KPS) [Count of Participants; unit: Participants] — 'Karnofsky Performance Status' (KPS) scale: 100 = Normal; no complaints; no evidence of disease; 90 = Able to carry on normal activity; minor signs or symptoms of disease; 80 = Normal activity with effort; some sign or symptoms of disease; 70 = Cares for self; unable to carry on normal activity or do active work.
  Participants
    100 | 0
    90 | 4
    80 | 8
    70 | 3

OUTCOME MEASURES:

1. Primary Outcome: 3-Month Progression-Free Survival (PFS3)
Description: PFS3 is the proportion of patients remaining alive and progression-free at 3-months from study entry. Progressive disease was established based on Response Assessment in Neuro-Oncology (RANO) criteria. RANO criteria has 5 potential categories: Complete Response (CR), Partial Response (PR), Stable Disease (SD), Progressive disease (PD) and Unknown. CR: disappearance of all enhancing lesions, stable or improved non-enhancing lesions, and stable or improved clinically. PR: >= 50% decrease in sum of perpendicular diameters of all measurable enhancing lesions, no progression of non-measurable disease, stable or improved non-enhancing lesions, and stable or improved clinically. PD: >25% increase in sum of perpendicular diameters of all measurable enhancing lesions, significant increase of non-enhancing lesions, any new lesions, clear clinical deterioration, failure to return for evaluation due to death or deteriorating condition. SD: does not qualify for CR,PR or PD.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ponatinib
Number analyzed (Participants) | 15
Participants | 0

2. Secondary Outcome: Best Radiographic Response
Description: Radiographic response was established based on Response Assessment in Neuro-Oncology (RANO) criteria with 5 potential categories: Complete Response (CR), Partial Response (PR), Stable Disease (SD), Progressive disease (PD) and Unknown status.
Time Frame: Disease was assessed radiographically for response every 8 weeks, assessed up to 24 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Ponatinib
Number analyzed (Participants) | 15
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 2
  Progressive Disease | 10
  Unknown | 3

3. Secondary Outcome: Overall Survival (OS)
Description: OS based on Kaplan-Meier is defined as the time from study entry to death or date last known alive.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ponatinib
Number analyzed (Participants) | 15
days | 98 [56 to 257]

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS based on Kaplan-Meier is defined as the time from study entry to the earliest documentation of disease progression or death. Progressive disease was established based on Response Assessment in Neuro-Oncology (RANO) criteria.
Time Frame: 3 months
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ponatinib
Number analyzed (Participants) | 15
days | 28 [27 to 30]

ADVERSE EVENTS:
Time Frame: Assessed each treatment cycle (1 cycle = 28 days) from time of first dose and up to day 30 post-treatment. Treatment duration in cycles was a median (range) of 1 (0-3). Assessed an average of 60 days.
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with ponatinib study treatment-attribution of at least possibly and causing a hospitalization, deemed serious by the treating investigator or grade 5 events per CTCAE v4. Other AEs were defined as events with ponatinib study treatment-attribution of at least possibly and not requiring a hospitalization or deemed non-serious by treating investigator.
Arm/Group | Ponatinib
All-Cause Mortality (participants affected / at risk) | 4/15
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ponatinib (N=15)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) — Grade 2
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ponatinib (N=15)
Anemia (Blood and lymphatic system disorders) | 1 (1) — Grade 1
Abdominal Pain (Gastrointestinal disorders) | 1 (1) — Grade 1
Constipation (Gastrointestinal disorders) | 1 (1) — Grade 1
Constipation (Gastrointestinal disorders) | 2 (2) — Grade 2
Diarrhea (Gastrointestinal disorders) | 1 (1) — Grade 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) — Grade 1
Mucositis Oral (Gastrointestinal disorders) | 1 (1) — Grade 1
Pancreatitis (Gastrointestinal disorders) | 1 (1) — Grade 2
Fatigue (General disorders) | 4 (4) — Grade 1
Fatigue (General disorders) | 2 (2) — Grade 2
Fatigue (General disorders) | 3 (3) — Grade 3
Alanine aminotransferase increased (Investigations) | 3 (3) — Grade 1
Alkaline phosphatase increased (Investigations) | 2 (2) — Grade 1
Aspartate aminotransferase increased (Investigations) | 3 (3) — Grade 1
CD4 lymphocytes decreased (Investigations) | 1 (1) — Grade 2
GGT increased (Investigations) | 2 (2) — Grade 1
Lipase increased (Investigations) | 2 (2) — Grade 3
Lymphocyte count decreased (Investigations) | 1 (1) — Grade 3
Platelet count decreased (Investigations) | 1 (1) — Grade 1
Platelet count decreased (Investigations) | 4 (4) — Grade 2
Serum amylase increased (Investigations) | 1 (1) — Grade 1
Serum amylase increased (Investigations) | 1 (1) — Grade 2
Anorexia (Metabolism and nutrition disorders) | 2 (2) — Grade 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) — Grade 1
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) — Grade 1
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) — Grade 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) — Grade 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 1
Hypertension (Vascular disorders) | 2 (2) — Grade 2
Hypertension (Vascular disorders) | 2 (2) — Grade 3
Diarrhea (Gastrointestinal disorders) | 1 (1) — Grade 2
Nausea (Gastrointestinal disorders) | 1 (1) — Grade 1
Alanine aminotransferase increased (Investigations) | 1 (1) — Grade 3
Aspartate aminotransferase increased (Investigations) | 1 (1) — Grade 3
Constipation (Gastrointestinal disorders) | 1 (1) — Grade 3
Weight loss (Investigations) | 1 (1) — Grade 1
Anorexia (Metabolism and nutrition disorders) | 2 (2) — Grade 2
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 2
Other - Mucosal lesions (Metabolism and nutrition disorders) | 1 (1) — Grade 1
Other - rash (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 1
Dysgeusia (Nervous system disorders) | 1 (1) — Grade 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-15): https://cdn.clinicaltrials.gov/large-docs/64/NCT02478164/Prot_SAP_000.pdf